CLINICAL TRIAL: NCT04459871
Title: A Phase 3, Stratified Randomized, Double-blind, Placebo-controlled Study of Topical Recombinant Human Thrombin (rhThrombin) in Surgical Hemostasis
Brief Title: Safety and Efficacy of Topical Recombinant Human Thrombin(rhThrombin) for Surgical Hemostasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZGrhT002
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Surgical Hemostasis
Keywords: hepatic resection; rhThrombin,topical
MeSH Terms: interventions — recombinant human thrombin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): The topical recombinant human thrombin(rhThrombin) was prepared into 1000IU/mL solution with 10ml normal saline and used in combination with absorbable gelatin spongeat at appropriate bleeding evaluation site(s).
  Interventions: Biological: recombinant human Thrombin(CHO cell)
- The control group (Placebo Comparator): The placebo was prepared into a solution with 10mL normal saline and used in combination with absorbable gelatin sponge at appropriate bleeding evaluation site(s).
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: recombinant human Thrombin(CHO cell) — 2 rhThrombin, dissolved in 5mL sterile saline and mixed, the final solution contains 1000IU/mL rhThrombin solution (clear and transparent liquid).
  Other Names: rhThrombin
  Arms: The experimental group
Biological: placebo — placebo, dissolved in 5mL sterile saline and mixed, the final solution contains 1000IU/mL rhThrombin solution (clear and transparent liquid).
  Arms: The control group

SUMMARY:
A multicenter, stratified randomized, double-blind, placebo-controlled, phase 3 clinical trial.

DETAILED DESCRIPTION:
After establishing eligibility, subjects will be randomized in a 2:1 ratio to receive rhThrombin (1000 U/mL) or placebo. During a surgical procedure, study participants will be treated with blinded study drug (rhThrombin or placebo) in combination with an absorbable gelatin sponge at appropriate bleeding evaluation site(s). 510 patients will participate in the study.

In this study, stratified random enrollment was conducted according to the condition(experimental group or control group) of the subjects.Stratification factors were centered, gender (male/female) and age (18 ≤ age <60/60 ≤ age ≤70).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old (including 18 and 70 years old), male or female;
* Patients with wedge-shaped liver resection or anatomical liver resection(1-5 consecutive liver segments);
* After the operation was controlled by standard surgical hemostasis, there were still patients with mild/moderate bleeding lesions (bleeding, non-arterial bleeding);
* Electrolytes (K, Na, CL, Ca, P, Mg) and ECG are normal or abnormal, Investigators believe that patients who do not affect surgery
* No other therapeutic surgery within 4 weeks before enrollment;
* Patients who have not used blood products within 24 hours before surgery;
* In compliance with the requirements of the ethics committee, patients voluntarily signed informed consent and were able to conduct visits as required by the protocol.

Exclusion Criteria:

* Known diseases of the blood system, including patients with coagulopathy or bleeding tendency;
* Patients with unstable vital signs for more than 24 hours;
* A history of severe heart, brain, and vascular disease within 6 months, including patients with a history of TIA, non-disabling cerebral infarction, myocardial infarction, unstable angina, or intracranial hemorrhage;
* Active bleeding or abnormal coagulation function (PT>16s, APTT>43s, INR≥2) or receiving thrombolysis, anticoagulation or antiplatelet therapy;
* Have used drugs that affect the function of the coagulation system within 1 week before surgery (including but not limited to: aspirin, clopidogrel, ticlopidine, fensulfamide, desmopressin, aminotoluic acid, dipyridamole, ginkgo Leaf preparations, heparin, warfarin, citrate, hemagglutinin, Vk, anti-fibrotic solvents, hemostatic, Vc, etc.);
* Women during pregnancy and lactation;
* Participants who participated in clinical trials of other drugs within 4 weeks before enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
The rate of complete hemostasis within 6 minutes. | 6 minutes
  Those who did not stop bleeding within 6 minutes were defined as treatment failure.

SECONDARY OUTCOMES:
Incidence of adverse events(AE) | Up to 28 days
  An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment.
Time to Hemostasis(TTH) | Evaluate the effect of hemostasis every 30sec until hemostasis is completed or 6 minutes of observation is completed
  TTH will be assessed for up to 6 minutes
Immunogenicity | At baseline and Day 29
  Positive rate of anti-recombinant human thrombin neutralizing antibody.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Yan, PhD, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China